CLINICAL TRIAL: NCT06661031
Title: Developing a Telehealth + mHealth Cannabis Use Intervention for Young Adults
Acronym: CAN-DO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lydia Shrier, Research Director, Division of Adolescent/Young Adult Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00049240; 1R34DA060500-01A1 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cannabis Use Disorder
Keywords: cannabis use; behavioral intervention; young adult
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The oral fluid testing pilot is a single-arm preliminary examination of remote oral fluid test feasibility and acceptability (anticipated n = up to 5).
  The pilot randomized controlled trial is a parallel, 2-arm, trial with 1:1 randomized allocation to the MOMENT-V intervention versus Enhanced Care, stratified by sex (male vs. not male), race (Black or African American vs. not Black or African American), cannabis use frequency (daily vs. not daily), and site (Boston Children's Hospital Adolescent/Young Adult Medical Practice vs. Martha Eliot Health Center Adolescent Clinic) (anticipated n=60).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care arm (Other): Participants meet with a study counselor 1-on-1 via videoconference to review a brochure containing cannabis information and treatment resources.
  Interventions: Behavioral: Enhanced Usual Care
- Intervention arm (Experimental): Participants meet with a counselor 1-on-1 via videoconference and receive MOMENT-V (mHealth intervention involving 2 Motivational Enhancement Therapy [MET] sessions with a trained counselor and 2 weeks of smartphone-based Ecological Momentary Assessment [EMI]).
  Interventions: Behavioral: Motivational Enhancement Therapy plus Ecological Momentary Intervention
- Oral fluid test pilot (No Intervention): Prior to RCT, single-arm pilot to test feasibility and acceptability of remote oral fluid testing.

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy plus Ecological Momentary Intervention — Two Motivational Enhancement Therapy (MET) sessions (1st, ~45 minutes; 2nd, ~30 minutes) between counselor and participant occur one week apart. MET sessions are personalized, interactive, face-to-face, and delivered according to a manual. MET session discussion topics include triggers for cannabis use, life goals/values, and development of a change plan. Participants then complete a 2-week Ecological Momentary Intervention (EMI) period. Survey prompts are sent 4x/day (3x/day at quasi-randomized times, 1x/day at fixed time; ~2 mins each) that ask about the participant's recent cannabis use. Depending on answers reported, the participant can receive tailored messages that support their self-efficacy and prompt use of coping strategies.
  Other Names: MOMENT-V
  Arms: Intervention arm
Behavioral: Enhanced Usual Care — Participants meet with a study counselor 1-on-1 via videoconference to review a brochure containing cannabis information and treatment resources.
  Arms: Enhanced Usual Care arm

SUMMARY:
The goal of this clinical trial is to determine 1) feasibility of the MOMENT-V intervention for cannabis use disorder in young adults, 2) feasibility of conducting the trial remotely, and 3) whether the MOMENT-V intervention reduces cannabis use frequency and problems. Researchers will compare the MOMENT-V intervention to usual care enhanced by a counselor meeting.

Participants will either meet with a counselor two times and use an app on their phone for two weeks, or meet with a counselor briefly one time. All participants will be asked to complete electronic surveys, interviews with a research assistant, and saliva drug testing at home over three months.

ELIGIBILITY:
For the oral fluid testing pilot

Inclusion Criteria:

* Primary care patient of the Boston Children's Hospital Adolescent/Young Adult Medicine Practice
* Participation in MOMENT-V open pilot
* Ownership of a smartphone
* Availability for the 2-week study duration

Exclusion Criteria:

* Inability/Unwillingness to provide contact information
* Current pregnancy or parenting

For the pilot RCT

Inclusion Criteria:

* Primary care patient of the Boston Children's Hospital Adolescent/Young Adult Medicine Practice or Martha Eliot Health Center Adolescent Clinic
* 18 to 26 years old
* Cannabis Use Disorders Identification Test-Revised (CUDIT-R) score of ≥12
* Recreational cannabis use on >3 days/week, on average, in the past 30 days
* Ownership of a smartphone that is PIN- or password-protected
* Ability to read and speak English
* Availability for the 6-month study duration

Exclusion Criteria:

* Inability/Unwillingness to provide contact information
* Written certification from a physician for marijuana for medical use
* Current participation in a substance use treatment program or research study
* Current pregnancy or parenting
* Participation in prior MOMENT or MOMENT-V research

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Intervention completion | At week 3 (Upon completion of 2-week EMI period)
  [Aim 1] Percent of participants assigned to the intervention arm completing the intervention (defined as both MET sessions and any EMI surveys). Benchmark: ≥80%
EMI engagement | In weeks 1-3 (during 2-week EMI period)
  [Aim 1] Percent of days on which participant responded to at least one survey during the 14 days of EMI. Benchmark: Median of ≥80% across intervention participants
Acceptability: Overall satisfaction | At 6-month timepoint
  [Aim 1] Satisfaction with intervention measured on the Client Satisfaction Questionnaire-8, an 8-item 4-point scale on which scores range from 8-32, with higher scores indicating greater satisfaction.
  Benchmark: ≥80% of participants with a scale score ≥24 (mean item score of ≥3 out 4)
Acceptability: Components | At week 0, week 1, and week 3
  [Aim 1] Measure of acceptability (usability, likability, perceived effect, burden) for each intervention component (2 MET sessions and EMI). Components assessed with an 11- or 12-item 5-point Likert-type scales (1, Strongly Disagree to 5, Strongly Agree) developed for the study. Higher scores indicate greater acceptability.
  Benchmark for each scale: ≥80% of participants with mean item score ≥4 out of 5
Screening | During recruitment (upon completion of eligibility survey: pre-enrollment, pre-Baseline)
  [Aim 2] Number of patients self-screening per month. Benchmark: ≥13 per month
Eligibility | During recruitment (upon completion of eligibility survey: pre-enrollment, pre-Baseline)
  [Aim 2] Number of patients eligible per month. Benchmark: ≥6 per month
Enrollment | Upon enrollment
  [Aim 2] Number of patients enrolled per month. Benchmark: ≥3 per month
Retention in trial | At 3-week timepoint, 3-month timepoint, 6-month timepoint
  [Aim 2] Percent of participants retained at each assessment time point (3 weeks, 3 months, 6 months, by assigned condition.
  Benchmark: ≥80% at each time point
Days of cannabis use | At Baseline, 3-week timepoint, 3-month timepoint, 6-month timepoint
  [Aim 3] Number of cannabis use days measured on Timeline Follow-Back (TLFB) calendar
Times of cannabis use | At Baseline, 3-week timepoint, 3-month timepoint, 6-month timepoint
  [Aim 3] Number of cannabis use times measured on TLFB calendar
Negative consequences of cannabis use | At Baseline, 3-month timepoint, 6-month timepoint
  [Aim 3] Number of negative consequences (problems) measured on the 19-item Marijuana Problems Scale

SECONDARY OUTCOMES:
Therapeutic alliance | At week 1
  [Aim 1] Working Alliance Inventory - Short Form, 12-items, 5-point Likert-type scale, total scale score and subscale scores (affective bond, perceived agreement on tasks, perceived agreement on goals; 4 items each), participant ("client") and observer versions reported separately and tested for agreement.
  Benchmark: ≥80% of participants with total score ≥48 (mean item score ≥4), participant version
MET counselor adherence to MI principles | At week 0 and week 1
  [Aim 1] Measure of counselor adherence to MI principles in each MET session, as reported by participant. Sessions assessed with 7- to 9-item 5-point Likert-type scales (Strongly Disagree to Strongly Agree) developed for the study.
  Benchmark for each scale: ≥80% of participants with mean item score ≥4 out of 5
Duration of study activities | All timepoints, upon completion of each timepoint (Baseline, week 0, week 1, weeks 1-3 [two-week EMI period], 3-weeks, 3-months, 6-months)
  [Aim 2] Duration of each study activity (in minutes)
Cannabis use disorder (CUD) symptoms | At Baseline, 3-month timepoint, 6-month timepoint
  [Aim 3] Symptom count measured by the Composite International Diagnostic Interview - Substance Abuse Module (CIDI-SAM)
Amount of THC used | At Baseline, 3-week timepoint, 3-month timepoint, 6-month timepoint
  [Aim 3] Number of standard THC units (1 unit = 5 mg THC) derived from number of familiar units (joints, vapes, gummies, etc.) x amount per unit (grams, milligrams, or milliliters) x estimated potency (% THC), measured on TLFB calendar.
  If unable to calculate standard THC units: Number of familiar units (joints, vapes, gummies, etc.)
Motivation to change cannabis use | At Baseline, week 0, week 1, 3-months, 6-months
  [Aim 3] One item each assessing readiness to, importance of, and confidence to change cannabis use, developed and used in our prior research, 11-point Likert-type scale for each. On follow-up, modified items about maintaining behavior if participant reports having started to change behavior but not having achieved change goals, or having changed behavior and achieved goals.
Psychological distress | At Baseline, 3-month timepoint, 6-month timepoint
  [Aim 3] Kessler Psychological Scale-6 (K6), assessing frequency of experiencing 6 symptoms in the past month on a 5-point Likert-type scale, with coding such that high scores indicate greater psychological distress.
Cognitive function | At Baseline, 3-month timepoint, 6-month timepoint
  [Aim 3] PROMIS Cognitive Function v.2.0 - Short Form 6a, 6 items, 5-point Likert-type response, measures participant-perceived cognitive deficits in the past 7 days. Age- and gender-weighted T scores, higher T-scores indicating better cognitive function.
Quality of life | At Baseline, 3-month timepoint, 6-month timepoint
  [Aim 3] PROMIS Global Health v1.2, a 10-item, 5-point Likert-type response (except pain item 0-10), participant-reported measure of physical, mental, and social health, in general except for past 7 days for emotional problems, fatigue, and pain. Age- and gender-weighted T scores, higher T-scores indicating better quality of life.

OTHER OUTCOMES:
Oral fluid acceptability | At 2-week timepoint in oral fluid pilot phase; At 3-month timepoint and 6-month timepoint in pilot RCT phase
  [Exploratory Aim] Measure of acceptability (usability, likability, burden), 5 items, 5-point Likert-type scale (1, Strongly Disagree to 5, Strongly Agree), with higher scores indicating greater acceptability
Oral fluid collection | For 3 days before and on the day of 2-week timepoint in oral fluid pilot phase; For 3 days before and on the day of 3-month timepoint and at 6-month timepoint in pilot RCT phase
  [Exploratory Aim] Number and percent of videos of self-testing completed out of those expected, per participant Number and percent of observations of self-testing during study visit out of those expected, per participant
Oral fluid - self-reported cannabis use agreement | For 3 days before and on the day of 2-week timepoint in oral fluid pilot phase; For 3 days before and on the day of 3-month timepoint and at 6-month timepoint in pilot RCT phase
  [Exploratory Aim] Agreement between oral fluid test results (positive/negative) and cannabis use reported on TLFB calendar for the day of testing or the day before testing (use/no use on either day)
Cannabis nonuse interval | For 4 days before and on the day of 2-week timepoint in oral fluid pilot phase; For 4 days before and on the day of 3-month timepoint and at 6-month timepoint in pilot RCT phase
  [Exploratory Aim] Oral fluid test results for delta-9-tetrahydrocannabinol on 4 consecutive days (all negative = nonuse over 5 days/any positive = use within the 5 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified survey and oral fluid testing data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified scientific data will be shared as soon as possible. De-identified scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: De-identified scientific data and metadata arising from the project will be archived in the openICPSR repository. De-identified scientific data from this project will be findable through summary information (metadata) that will be readily available on the Center for Adolescent Behavioral Health Research website, the repository website, and clinicaltrials.gov.

REFERENCES:
- [Background] Shrier LA, Rhoads A, Burke P, Walls C, Blood EA. Real-time, contextual intervention using mobile technology to reduce marijuana use among youth: a pilot study. Addict Behav. 2014 Jan;39(1):173-80. doi: 10.1016/j.addbeh.2013.09.028. Epub 2013 Oct 4. PMID 24139665
- [Background] Shrier LA, Burke PJ, Kells M, Scherer EA, Sarda V, Jonestrask C, Xuan Z, Harris SK. Pilot randomized trial of MOMENT, a motivational counseling-plus-ecological momentary intervention to reduce marijuana use in youth. Mhealth. 2018 Jul 30;4:29. doi: 10.21037/mhealth.2018.07.04. eCollection 2018. PMID 30148142
- [Background] Shrier LA, McCaskill NH, Smith MC, O'Connell MM, Gluskin BS, Parker S, Everett V, Burke PJ, Harris SK. Telehealth counseling plus mHealth intervention for cannabis use in emerging adults: Development and a remote open pilot trial. J Subst Use Addict Treat. 2024 Nov;166:209472. doi: 10.1016/j.josat.2024.209472. Epub 2024 Aug 5. PMID 39111371